CLINICAL TRIAL: NCT03251924
Title: A Phase 1/2 Dose Escalation and Combination Cohort Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Efficacy of BMS-986226 Alone or in Combination With Nivolumab or Ipilimumab in Patients With Advanced Solid Tumors
Brief Title: A Dose Escalation and Combination Immunotherapy Study to Evaluate BMS-986226 Alone or in Combination With Nivolumab or Ipilimumab in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study CA021-002 was terminated because the Sponsor discontinued further development of BMS-986226 due to a change in business objectives. The decision for the study closure was not related to any safety concerns associated with BMS-986226.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA021-002; 2017-000238-73 (EudraCT Number)
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Cancer; Tumors; Neoplasm; Malignancy
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; Ipilimumab; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986226 (Experimental): administered intravenously
  Interventions: Drug: BMS-986226; Biological: Tetanus Vaccine
- BMS-986226 and Nivolumab (Experimental): administered intravenously
  Interventions: Drug: BMS-986226; Biological: Nivolumab; Biological: Tetanus Vaccine
- BMS-986226 and Ipilimumab (Experimental): administered intravenously
  Interventions: Drug: BMS-986226; Biological: Ipilimumab; Biological: Tetanus Vaccine

INTERVENTIONS:
Drug: BMS-986226 — specified dose on specified days
Biological: Nivolumab — specified dose on specified days
  Other Names: BMS-936558; PD-1 receptor blocking monoclonal antibody [mAb]; Opdivo
  Arms: BMS-986226 and Nivolumab
Biological: Ipilimumab — specified dose on specified days
  Other Names: BMS-734016; MDX010; Checkpoint blocking antibody that recognizes CTLA-4; Yervoy
  Arms: BMS-986226 and Ipilimumab
Biological: Tetanus Vaccine — specified dose on specified days

SUMMARY:
The purpose of this study is to investigate BMS-986226 administered alone or in combination with nivolumab or ipilimumab.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Advanced solid tumors
* Histological or cytological confirmation of a malignancy that is advanced (metastatic and/or unresectable) with measureable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or PCWG3 (prostate only).
* At least 1 lesion accessible for biopsy in addition to the target lesion
* Participants must have received, and then progressed or been intolerant to, at least 1 standard treatment regimen
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Exclusion Criteria:

* Participants with active central nervous system (CNS) metastases, untreated CNS metastases, or with the CNS as the only site of disease are excluded (controlled brain metastases will be allowed to enroll)
* Participants with carcinomatous meningitis
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Active, known, or suspected autoimmune disease
* Uncontrolled or significant cardiovascular disease
* Participants with known allergies to egg products, neomycin and tetanus toxoid.
* Prior adverse reaction to tetanus toxoid- containing vaccines.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (5):
  - Local Institution - 0005, Boston, Massachusetts
  - Local Institution - 0012, St Louis, Missouri
  - Local Institution - 0002, Hackensack, New Jersey
  - Local Institution - 0001, Philadelphia, Pennsylvania
  - Local Institution - 0004, Nashville, Tennessee
- Canada (3):
  - Local Institution - 0014, Edmonton, Alberta
  - Local Institution - 0006, Hamilton, Ontario
  - Local Institution - 0003, Toronto, Ontario
- Spain (2):
  - Local Institution - 0007, Madrid
  - Local Institution - 0008, Madrid
- Switzerland (3):
  - Local Institution - 0009, Chur
  - Local Institution - 0010, Lausanne
  - Local Institution - 0011, Zurich

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were treated with BMS-986226 in combination with nivolumab (Parts B1 and B2) and no participants were treated in Parts D and E
Groups:
- Preliminary - BMS-986226 2 mg: Preliminary safety cohort participants received BMS-986226 2 mg every 4 weeks
- Preliminary - BMS-986226 8 mg: Preliminary safety cohort participants received BMS-986226 8 mg every 4 weeks
- Part A - BMS-986226 25 mg: Part A cohort participants received BMS-986226 25 mg every 4 weeks for 24 weeks
- Part A - BMS-986226 80 mg: Part A cohort participants received BMS-986226 80 mg every 4 weeks for 24 weeks
- Part A - BMS-986226 200 mg: Part A cohort participants received BMS-986226 200 mg every 4 weeks for 24 weeks
- Part A - BMS-986226 400 mg: Part A cohort participants received BMS-986226 400 mg every 4 weeks for 24 weeks
- Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg: Part C1 cohort participants received BMS-986226 25 mg every 12 weeks plus Ipilimumab 3 mg/kg every 4 weeks
- Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg: Part C1 cohort participants received BMS-986226 200 mg every 12 weeks plus Ipilimumab 3 mg/kg every 4 weeks
- Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg: Part C2 cohort participants received BMS-986226 25 mg every 4 weeks plus Ipilimumab 3 mg/kg every 4 weeks
Period: Overall Study
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Started | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Not Completed | 6 | 7 | 7 | 11 | 9 | 9 | 7 | 11 | 8
Not completed — Disease Progression | 6 | 6 | 7 | 8 | 8 | 7 | 6 | 10 | 6
Not completed — Adverse Event unrelated to study drug | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Study Drug Toxicity | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant request to discontinue study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Total
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (10.4) | 58.3 (7.8) | 63.6 (12.3) | 62.5 (9.7) | 55.3 (15.9) | 61.7 (16.9) | 55.7 (9.6) | 62.3 (11.7) | 58.3 (7.1) | 59.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 5 | 3 | 3 | 4 | 5 | 2 | 28
  Male | 5 | 5 | 4 | 6 | 6 | 6 | 6 | 7 | 7 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 5 | 5 | 4 | 5 | 4 | 2 | 6 | 8 | 5 | 44
  Unknown or Not Reported | 0 | 1 | 2 | 6 | 5 | 6 | 3 | 4 | 3 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  White | 4 | 6 | 6 | 10 | 9 | 9 | 7 | 12 | 6 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose up to 100 days post last dose, up to approximately 31 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9

2. Primary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose up to 100 days post last dose, up to approximately 31 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants | 2 | 3 | 2 | 10 | 5 | 9 | 5 | 9 | 5

3. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Meeting Dose Limiting Toxicity (DLT) Criteria
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Dose limiting toxicity (DLT) is defined based on the incidence, intensity, and duration of AEs for which no clear alternative cause is identified. The DLT period will be 28 days (4 weeks) in the Preliminary Safety Cohorts. Any toxicities that occur beyond the 4-week DLT period will also be considered in dose-level decisions. For the purpose of participant management, any AE that meets DLT criteria, regardless of the cycle in which it occurs, will lead to discontinuation of study treatment. AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Time Frame: From first dose up to 100 days post last dose, up to approximately 31 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: The Number of Participants Experiencing Adverse Events Leading to Discontinuation
Description: as for outcome 1
Time Frame: From first dose up to 100 days post last dose, up to approximately 31 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 3 | 2

5. Primary Outcome: The Number of Participants Experiencing Adverse Events Resulting in Death
Description: as for outcome 1
Time Frame: From first dose up to 100 days post last dose, up to approximately 31 months
Population: All treated paricipants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants | 5 | 3 | 5 | 8 | 5 | 7 | 7 | 8 | 5

6. Primary Outcome: The Number of Participants Experiencing Clinical Laboratory Abnormalities
Description: The number of participants experiencing abnormal laboratory results of Grade 3 or higher. Laboratory values will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 with Grade 3=severe and Grade 4=life threatening.
Time Frame: From first dose up to 30 days post last dose (approximately 28 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Participants
  HEMOGLOBIN | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
  LYMPHOCYTES (ABSOLUTE) | 0 | 1 | 1 | 3 | 2 | 3 | 2 | 4 | 3
  LYMPHOCYTES (RELATIVE) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  ALKALINE PHOSPHATASE | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 2 | 0
  ASPARTATE AMINOTRANSFERASE | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
  ALANINE AMINOTRANSFERASE | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  G-GLUTAMYL TRANSFERASE | 1 | 2 | 1 | 4 | 3 | 2 | 6 | 3 | 1
  BILIRUBIN, TOTAL | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  PHOSPHATE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  LIPASE, TOTAL | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1
  HYPONATREMIA | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  HYPERKALEMIA | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HYPERGLYCEMIA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOKALEMIA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of all treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) as assessed by investigator per RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must also have reduction in the short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. BOR for a participant is defined as the best response designation recorded between the date of first dose (or date of randomization) and the date of first objectively documented progression per RECIST 1.1 or the date of subsequent therapy, whichever occurs first.
Time Frame: From first dose up to documented disease progression, up to 48 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 9 | 9 | 9 | 10 | 12 | 9
Percentage of participants | 0 [0.0 to 45.9] | 0 [0.0 to 41.0] | 0 [0.0 to 41.0] | 0 [0.0 to 28.5] | 0 [0.0 to 33.6] | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 8.3 [0.2 to 38.5] | 0 [0.0 to 33.6]

8. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR for a participant with confirmed response is defined as the time from the date of first response CR or PR to the date of first objectively documented tumor progression as determined using RECIST v1.1 or death due to any cause, whichever occurs first. Participant who remain alive and have not progressed will be censored on the date of their last tumor assessment. Participants who started subsequent anticancer therapy without a prior reported progression will be censored at the last tumor assessment prior to initiation of the subsequent anticancer therapy. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must also have reduction in the short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to the date of the first objectively documented tumor progression or death, whichever occurs first (up to approximately 24 months)
Population: All treated participants with complete response (CR) or partial response (PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Months |  |  |  |  |  |  |  | NA [23.4 to 23.4] — Median not calculable because data were only collected for 1 participant. |

9. Secondary Outcome: Progression Free Survival (PFS) Rate at 24 Weeks
Description: The PFSR is defined as the Kaplan Meier estimate of percentage of treated participants remaining progression free and surviving at the prespecified timepoint of 24 weeks since the first dosing date. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of 1 or more new lesions is also considered progression.)
Time Frame: At 24 weeks
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7 | 11 | 9 | 9 | 10 | 12 | 9
Percentage of participants | 16.7 [0.8 to 51.7] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 8.3 [0.5 to 31.1] | 18.8 [1.1 to 53.5]

10. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) for BMS-986226
Description: ADA for BMS-986226 is defined as the number of participants found to have seroconverted or boosted their pre-existing ADA during the study period. Baseline ADA positive is defined as ADA is detected in the last sample before initiation of treatment. ADA positive is defined as 1) an ADA detected (positive seroconversion) sample in a participant for whom ADA is not detected at baseline, or (2) an ADA detected sample with ADA titer to be at least 4-fold or greater (≥) than baseline positive titer.
Time Frame: Predose on cycles 1-6, post dose on C1D15, and 30, 60, and 100 days post last dose (up to approximately 31 months)
Population: All treated participants with baseline and at lease one post-baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 11 | 9 | 8 | 8 | 11 | 9
Participants
  Baseline ADA Positive | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  ADA Positive after initiation of treatment | 4 | 6 | 3 | 8 | 4 | 4 | 8 | 9 | 8

11. Secondary Outcome: Changes From Baseline in Cell Surface ICOS Expression on T Cells
Description: Summary measures of changes in Median of Fluorescence of ICOS (MFI) from baseline to the last evaluable time point in cell surface Inducible Costimulator (ICOS) expression on T cells. Baseline = last non missing value prior or on to the first dosing. MFI is a unit for median fluorescence intensity. This unit allows for measurement of relative expression of cell surface markers by a flow cytometer. For the ICOS expression assay, whole blood samples collected from patients on study were incubated with fluorescently labeled antibodies that specifically bind to ICOS. Samples were then analyzed for changes in MFI by flow cytometry. An increase in MFI between patient samples corresponds to an increase in cell surface ICOS expression on target cell subsets.
Time Frame: From baseline up to pre-dose and 4 hours post dose on C1D1 and pre-dose and 4 hours post dose on C2D1 (approximately 31 months)
Population: Biomarker Evaluable Participants: All treated participants with available biomarker data
Measure: Median (Full Range); unit: Median of Fluorescence of ICOS (MFI)
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 4 | 6 | 7 | 10 | 8 | 9 | 9 | 10 | 6
Median of Fluorescence of ICOS (MFI)
  Baseline Response | 985.5 [554 to 1243] | 659.0 [455 to 775] | 878.0 [599 to 1361] | 482 [197 to 912] | 434.0 [169 to 884] | 634.0 [94 to 1166] | 592.0 [162 to 933] | 714.0 [234 to 1438] | 506.5 [20 to 943]
  C1D1- Pre-Dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0
  C1D1- Pre-Dose | -394.0 [-394 to 394] |  |  |  |  | -636.0 [-636 to -636] |  |  |
  C1D1- 4 hours post dose: number analyzed (Participants) | 1 | 6 | 5 | 5 | 4 | 7 | 2 | 10 | 5
  C1D1- 4 hours post dose | -1049.0 [-1049 to -1049] | -603.0 [-603 to -603] | -762.0 [-847 to -565] | -391.0 [-635 to -176] | -324.0 [-481 to -95] | -545.0 [-1029 to -184] | -382.5 [-649 to -116] | -654.5 [-1405 to -214] | -490.0 [-928 to -429]
  C2D1- Pre-Dose: number analyzed (Participants) | 3 | 4 | 5 | 6 | 5 | 2 | 7 | 8 | 4
  C2D1- Pre-Dose | -421.0 [-729 to -31] | -26.0 [-538 to 104] | -414.0 [-1101 to 630] | -153.0 [-774 to -38] | -185.0 [-865 to -177] | -627.0 [-632 to -622] | -294.0 [-500 to 308] | -185.5 [-1155 to 430] | 11.5 [-104 to 148]
  C2D1- 4 hours post dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 4
  C2D1- 4 hours post dose |  |  |  | -167.5 [-229 to -106] | -336.5 [-507 to -166] | -567.0 [-615 to -372] |  |  | -465.5 [-911 to 254]

12. Secondary Outcome: Changes From Baseline in ICOS Ligand+ B Cells
Description: Summary measures of changes in Median of Fluorescence of ICOS (MFI) from baseline to the last evaluable time point in ICOS ligand+ B cells in the tumor and peripheral blood. Baseline = last non missing value prior or on to the first dosing. MFI is a unit for median fluorescence intensity. This unit allows for measurement of relative expression of cell surface markers by a flow cytometer. For the ICOS expression assay, whole blood samples collected from patients on study were incubated with fluorescently labeled antibodies that specifically bind to ICOS. Samples were then analyzed for changes in MFI by flow cytometry. An increase in MFI between patient samples corresponds to an increase in cell surface ICOS expression on target cell subsets.
Time Frame: From baseline up to pre-dose and 4 hours post dose on C1D1, 72 hours post dose on C1D4, and pre-dose on C2D1 (approximately 31 months)
Population: Biomarker Evaluable Participants: All treated participants with available biomarker data
Measure: Median (Full Range); unit: Median of Fluorescence of ICOS (MFI)
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 4 | 6 | 6 | 10 | 8 | 9 | 9 | 10 | 8
Median of Fluorescence of ICOS (MFI)
  Baseline Response | -9.0 [-94 to 185] | -33.0 [-70 to 67] | 2.5 [-99 to 95] | 40.5 [-90 to 127] | -60.5 [-171 to 74] | 57.0 [-100 to 182] | -15.0 [-79 to 70] | -11.5 [-113 to 41] | 39.0 [-56 to 103]
  C1D1 - 4 hours post dose: number analyzed (Participants) | 1 | 1 | 4 | 5 | 4 | 8 | 2 | 10 | 7
  C1D1 - 4 hours post dose | -106.0 [-106 to -106] | -2.0 [-2 to -2] | -3.0 [-48 to 37] | 1.0 [-9 to 23] | -13.5 [-55 to 0] | 9.5 [-16 to 99] | 3.5 [1 to 6] | 0.0 [-14 to 37] | -6.0 [-21 to 40]
  C1D4- 72 hours post dose: number analyzed (Participants) | 3 | 4 | 5 | 9 | 8 | 9 | 2 | 10 | 8
  C1D4- 72 hours post dose | 11.0 [-181 to 58] | 102.0 [-28 to 190] | 170.0 [118 to 210] | 37.0 [-143 to 231] | 64.5 [-71 to 127] | 29.0 [-106 to 88] | 90.0 [17 to 163] | 70.0 [3 to 143] | 33.5 [-28 to 121]
  C2D1- Pre dose: number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 2 | 7 | 8 | 6
  C2D1- Pre dose | -4.0 [-267 to 54] | -24.0 [-211 to 24] | 96.0 [-167 to 207] | -17.0 [-100 to 170] | 103.5 [-39 to 216] | -28.0 [-74 to 18] | -9.0 [-129 to 83] | 61.5 [-20 to 186] | -17.0 [-175 to 103]

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is the maximum serum concentration that a drug achieves after the drug has been administered and before the administration of a second dose.
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 5 | 7 | 6 | 11 | 9 | 8 | 8 | 11 | 9
ng/mL
  C1D1 | 733 (NA) — Geometric Coefficient of Variation not calculated. %CV=37 | 2250 (NA) — Geometric Coefficient of Variation not calculated. %CV=20 | 6609 (NA) — Geometric Coefficient of Variation not calculated. %CV=23 | 19524 (NA) — Geometric Coefficient of Variation not calculated. %CV=28 | 41698 (NA) — Geometric Coefficient of Variation not calculated. %CV=33 | 85905 (NA) — Geometric Coefficient of Variation not calculated. %CV=37 | 5440 (NA) — Geometric Coefficient of Variation not calculated. %CV=35 | 43309 (NA) — Geometric Coefficient of Variation not calculated. %CV=28 | 3451 (NA) — Geometric Coefficient of Variation not calculated. %CV=53
  C2D1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 5 | 5 | 0 | 1 | 2
  C2D1 |  | 1050 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 7220 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 23322 (NA) — Geometric Coefficient of Variation not calculated. %CV=16 | 45054 (NA) — Geometric Coefficient of Variation not calculated. %CV=36 | 91931 (NA) — Geometric Coefficient of Variation not calculated. %CV=108 |  | 30200 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 2697 (NA) — Geometric Coefficient of Variation not calculated. %CV=7
  C3D1: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1
  C3D1 |  | 1060 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 3168 (NA) — Geometric Coefficient of Variation not calculated. %CV=12 | 15000 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 41700 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 76700 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  | 3880 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses.

14. Secondary Outcome: Effective Elimination Half-Life (T-HALFeff)
Description: Effective elimination half-life that explains the degree of accumulation observed
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C2D1 and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hours
  C2D1 |  |  |  | 212 (9.4) | 102 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  |  |  |
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  C3D1 |  |  |  |  | 308 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  |  |  |

15. Secondary Outcome: Trough Observed Serum Concentrations (Ctrough)
Description: Trough observed serum concentrations (Ctrough) is defined as the concentration reached by a drug immediately before the next dose is administered
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C2D1 and C3D1. Pre-dose and 0.5 post dose on C4D1. Pre-dose on C5D1 and C6D1. Pre-dose and 0.5 hours post dose on C7D1. (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 5 | 4 | 1 | 1 | 1
ng/mL
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 5 | 4 | 1 | 0 | 1
  Cycle 2 Day 1 |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 27.0 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 943 (584.4) | 1501 (1202.9) | 1491 (1287.3) | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses.
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1
  Cycle 3 Day 1 |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 27.2 (20.72) | 892 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 180 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 3150 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses.
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1
  Cycle 4 Day 1 | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 504 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 800 (401.1) |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses.
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Cycle 5 Day 1 | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  |  |  | 3300 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  |  |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses.
  Cycle 6 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 6 Day 1 | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. |  |  |  |  |  |  |  |
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 7 Day 1 |  |  |  |  |  |  |  | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses. | 12.5 (NA) — Standard deviation not calculated due to insufficient number of participants with evaluable responses.

16. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Tmax is defined as the amount of time that a drug is present at the maximum concentration in serum
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Median (Full Range); unit: Hours
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 6 | 7 | 6 | 11 | 9 | 8 | 8 | 11 | 9
Hours
  C1D1: number analyzed (Participants) | 5 | 7 | 6 | 11 | 9 | 8 | 8 | 11 | 9
  C1D1 | 4.00 [0.067 to 4.22] | 0.283 [0.133 to 4.00] | 0.534 [0.467 to 4.50] | 1.25 [0.467 to 21.7] | 3.88 [0.467 to 24.0] | 4.00 [0.500 to 24.0] | 2.88 [0.467 to 4.50] | 1.02 [0.483 to 18.9] | 0.600 [0.467 to 22.0]
  C2D1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 5 | 5 | 0 | 1 | 2
  C2D1 |  | 0.600 [0.600 to 0.600] | 0.967 [0.967 to 0.967] | 4.00 [0.483 to 4.00] | 1.00 [0.433 to 4.52] | 4.00 [0.383 to 4.00] |  | 2.83 [2.83 to 2.83] | 2.24 [0.483 to 4.00]
  C3D1: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1
  C3D1 |  | 0.133 [0.133 to 0.133] | 0.534 [0.517 to 0.550] | 0.467 [0.467 to 0.467] | 1.03 [1.03 to 1.03] | 0.967 [0.967 to 0.967] |  |  | 0.500 [0.500 to 0.500]

17. Secondary Outcome: Area Under Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration [AUC (0-T)]
Description: AUC(0-t) (partial AUC) is defined as the area under the concentration-time curve from dosing (time 0) to time t. AUC(0-t) may be computed for one or more values of t, with specific values of t determined after observing the data.
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 5 | 7 | 6 | 11 | 9 | 8 | 8 | 11 | 9
h*ng/mL
  C1D1 | 33704 (NA) — Geometric Coefficient of Variation not calculated. %CV=12 | 175228 (NA) — Geometric Coefficient of Variation not calculated. %CV=33 | 682168 (NA) — Geometric Coefficient of Variation not calculated. %CV=23 | 1951486 (NA) — Geometric Coefficient of Variation not calculated. %CV=52 | 4966612 (NA) — Geometric Coefficient of Variation not calculated. %CV=53 | 8346408 (NA) — Geometric Coefficient of Variation not calculated. %CV=25 | 370356 (NA) — Geometric Coefficient of Variation not calculated. %CV=41 | 4805561 (NA) — Geometric Coefficient of Variation not calculated. %CV=60 | 277927 (NA) — Geometric Coefficient of Variation not calculated. %CV=54
  C2D1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 5 | 5 | 0 | 1 | 2
  C2D1 |  | 13921 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 933038 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 3534177 (NA) — Geometric Coefficient of Variation not calculated. %CV=14 | 5887547 (NA) — Geometric Coefficient of Variation not calculated. %CV=45 | 4070442 (NA) — Geometric Coefficient of Variation not calculated. %CV=60 |  | 2528949 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 35464 (NA) — Geometric Coefficient of Variation not calculated. %CV=39
  C3D1: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1
  C3D1 |  | 18442 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 81982 (NA) — Geometric Coefficient of Variation not calculated. %CV=128 | 2727643 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 5157593 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 7511434 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  | 55178 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses.

18. Secondary Outcome: Area Under the Concentration-Time Curve in 1 Dosing Interval [AUC (TAU)]
Description: AUC (TAU) is defined as the area under the plasma concentration-time curve from time zero to the end of the dosing interval
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 5 | 7 | 6 | 11 | 9 | 8 | 8 | 11 | 9
h*ng/mL
  C1D1 | 37392 (NA) — Geometric Coefficient of Variation not calculated. %CV=18 | 189031 (NA) — Geometric Coefficient of Variation not calculated. %CV=32 | 704072 (NA) — Geometric Coefficient of Variation not calculated. %CV=22 | 1992589 (NA) — Geometric Coefficient of Variation not calculated. %CV=51 | 5148217 (NA) — Geometric Coefficient of Variation not calculated. %CV=51 | 8740936 (NA) — Geometric Coefficient of Variation not calculated. %CV=26 | 404651 (NA) — Geometric Coefficient of Variation not calculated. %CV=42 | 5006775 (NA) — Geometric Coefficient of Variation not calculated. %CV=67 | 301365 (NA) — Geometric Coefficient of Variation not calculated. %CV=53
  C2D1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 2 | 0 | 0 | 0
  C2D1 |  |  | 933038 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 3693517 (NA) — Geometric Coefficient of Variation not calculated. %CV=12 | 5766681 (NA) — Geometric Coefficient of Variation not calculated. %CV=55 | 10833374 (NA) — Geometric Coefficient of Variation not calculated. %CV=4 |  |  |
  C3D1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  C3D1 |  | 19007 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 373429 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 2727643 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 5157593 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |  |

19. Secondary Outcome: Total Body Clearance (CLT)
Description: CLT is defined as the elimination of the drug from the body
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 3 | 4 | 2 | 0 | 0 | 0
mL/h
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 2 | 0 | 0 | 0
  C2D1 |  |  | 26.8 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 21.7 (NA) — Geometric Coefficient of Variation not calculated. %CV=13 | 34.7 (NA) — Geometric Coefficient of Variation not calculated. %CV=59 | 36.9 (NA) — Geometric Coefficient of Variation not calculated. %CV=4 |  |  |
  C3D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  C3D1 |  | 421 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  | 29.3 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 38.8 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |  |

20. Secondary Outcome: Average Concentration Over a Dosing Interval (Css-avg)
Description: Css-avg is defined as the average concentration over a dosing interval (AUC[TAU]/tau)
  Note: Coefficient of variation is reported in lieu of geometric coefficient of variation
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 3 | 4 | 2 | 0 | 0 | 0
ng/mL
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 2 | 0 | 0 | 0
  C2D1 |  |  | 1397 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 5499 (NA) — Geometric Coefficient of Variation not calculated. %CV=12 | 8581 (NA) — Geometric Coefficient of Variation not calculated. %CV=55 | 16115 (NA) — Geometric Coefficient of Variation not calculated. %CV=4 |  |  |
  C3D1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  C3D1 |  | 28.3 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 556 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 4065 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 7666 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |  |

21. Secondary Outcome: Accumulation Index - Area Under Curve (AI-AUC)
Description: Accumulation Index is defined as the extent of drug accumulation and determined by the ratio of plasma concentration at plateau over plasma concentration after the first dose. The area under curve is defined as the area under the plot of plasma concentration of a drug versus time after dosage which reflects the extent of exposure to a drug and its clearance rate from the body.
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1, and C3D1 (approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 3 | 4 | 1 | 0 | 0 | 0
Ratio
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 1 | 0 | 0 | 0
  C2D1 |  |  |  | 1.07 (NA) — Geometric Coefficient of Variation not calculated. %CV=9 | 0.856 (NA) — Geometric Coefficient of Variation not calculated. %CV=14 | 0.953 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |
  C3D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  C3D1 |  | 0.100 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  | 0.808 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 1.28 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |  |

22. Secondary Outcome: Accumulation Index - Cmax (AI-Cmax)
Description: Accumulation Index is defined as the extent of drug accumulation and determined by the ratio of plasma concentration at plateau over plasma concentration after the first dose. Cmax is the maximum serum concentration that a drug achieves after the drug has been administered and before the administration of a second dose.
Time Frame: Pre-dose, 0.5, 4, 24, 72, 168, 336, 504 hours post dose on C1D1, C2D1 and C3D1. Pre-dose and 0.5 post dose on C4D1. (Approximately 31 months)
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 3 | 5 | 4 | 0 | 1 | 2
Ratio
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1: number analyzed (Participants) | 0 | 1 | 0 | 3 | 5 | 4 | 0 | 0 | 2
  C2D1 |  | 0.475 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  | 1.19 (NA) — Geometric Coefficient of Variation not calculated. %CV=12 | 0.951 (NA) — Geometric Coefficient of Variation not calculated. %CV=5 | 0.861 (NA) — Geometric Coefficient of Variation not calculated. %CV=86 |  |  | 0.687 (23)
  C3D1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1
  C3D1 |  | 0.457 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 0.309 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 0.920 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 1.11 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 0.940 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  | 1.11 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses.
  C4D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  C4D1 |  |  |  |  |  |  |  | 0.633 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |

23. Secondary Outcome: Accumulation Index - Concentrations at the End of Dosing Interval (AI-CTAU)
Description: Accumulation Index is defined as the extent of drug accumulation and determined by the ratio of plasma concentration at plateau over plasma concentration after the first dose.
Time Frame: as for outcome 22
Population: Evaluable PK Population: All treated participants who have evaluable serum concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 3 | 4 | 1 | 0 | 0 | 0
Ratio
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 1 | 0 | 0 | 0
  C2D1 |  |  |  | 0.640 (NA) — Geometric Coefficient of Variation not calculated. %CV=10 | 1.12 (NA) — Geometric Coefficient of Variation not calculated. %CV=114 | 1.38 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |
  C3D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  C3D1 |  | NA (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  | 0.391 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. | 33.3 (NA) — Geometric Coefficient of Variation not calculated. %CV not calculated due to insufficient number of participants with evaluable responses. |  |  |  |
  C4D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 50 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 31 months)
Groups:
- Total: Total treated participants
Arm/Group | Preliminary - BMS-986226 2 mg | Preliminary - BMS-986226 8 mg | Part A - BMS-986226 25 mg | Part A - BMS-986226 80 mg | Part A - BMS-986226 200 mg | Part A - BMS-986226 400 mg | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg | Total
All-Cause Mortality (participants affected / at risk) | 5/6 | 3/7 | 5/7 | 8/11 | 5/9 | 7/9 | 7/10 | 8/12 | 5/9 | 53/80
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/7 | 2/7 | 10/11 | 5/9 | 9/9 | 5/10 | 9/12 | 5/9 | 50/80
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 7/7 | 10/11 | 9/9 | 9/9 | 10/10 | 12/12 | 9/9 | 79/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preliminary - BMS-986226 2 mg (N=6) | Preliminary - BMS-986226 8 mg (N=7) | Part A - BMS-986226 25 mg (N=7) | Part A - BMS-986226 80 mg (N=11) | Part A - BMS-986226 200 mg (N=9) | Part A - BMS-986226 400 mg (N=9) | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg (N=10) | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg (N=12) | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg (N=9) | Total (N=80)
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 5 | 4 | 6 | 5 | 6 | 4 | 33
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Assisted suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Preliminary - BMS-986226 2 mg (N=6) | Preliminary - BMS-986226 8 mg (N=7) | Part A - BMS-986226 25 mg (N=7) | Part A - BMS-986226 80 mg (N=11) | Part A - BMS-986226 200 mg (N=9) | Part A - BMS-986226 400 mg (N=9) | Part C1 - BMS-986226 25 mg + Ipilimumab 3 mg/kg (N=10) | Part C1 - BMS-986226 200 mg + Ipilimumab 3 mg/kg (N=12) | Part C2 - BMS-986226 25 mg + Ipilimumab 3 mg/kg (N=9) | Total (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1 | 3 | 2 | 4 | 0 | 14
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2 | 2 | 3 | 3 | 0 | 15
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0 | 4 | 1 | 1 | 0 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 6 | 3 | 3 | 0 | 16
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 4 | 3 | 14
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Fatigue (General disorders) | 2 | 1 | 1 | 4 | 3 | 5 | 3 | 5 | 1 | 25
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 6
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 4
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 1 | 0 | 10
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 5 | 8 | 8 | 4 | 6 | 3 | 40
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 6
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 2 | 1 | 0 | 4 | 3 | 1 | 15
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 8
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 6
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0 | 5 | 2 | 3 | 0 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 9
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Study CA021002 was terminated because the Sponsor discontinued further development of BMS-986226. The decision for the study closure was not related to any safety concerns associated with BMS-986226.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT03251924/Prot_SAP_000.pdf